CLINICAL TRIAL: NCT04340674
Title: Immediate Effects of a Telerehabilitation Program Based on Aerobic Exercise in Women With Fibromyalgia
Brief Title: Telerehabilitation Based on Aerobic Exercise in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Ignacio Hernando Garijo, Physiotherapist, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UValladolid
Record Dates: First submitted 2020-03-27; First posted 2020-04-09 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia
Keywords: exercise; aerobic exercise; telerehabilitation
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation based on aerobic exercise (Experimental): Aerobic low-impact exercise guided by audiovisual material. The intensity of exercise is adapted to each participant and is established according to the perceived effort after each session, according to the modified Borg perceived effort scale.
  Interventions: Other: Telerehabilitation based on aerobic exercise
- Control group (No Intervention): Group that maintain the same medical treatment and not receive additional intervention.

INTERVENTIONS:
Other: Telerehabilitation based on aerobic exercise — To perform different whole body aerobic exercises moderately intense according to Borg scale.
  Arms: Telerehabilitation based on aerobic exercise

SUMMARY:
Fibromyalgia syndrome is the most common cause of chronic generalized musculoskeletal pain and is characterized by pain associated with generalizad sensitivity, fatigue, sleep disturbances and psychological problems. Due to the chronic nature of the pathology and the great dependence on analgesic drugs that it often entails, in these patients it is considered necessary to provide an individualized approach and provide strategies that allow symptoms to be controlled conservatively and non-pharmacologically.

The objective of this trial is to analyse the immediate effects on pain, mechanical pain sensitivity, impact of fibromyalgia, pain catastrophizing, psychological distress and physical function when a telerehabilitation program based on aerobic exercise is applied in women with fibromyalgia.

For this purpose the investigators conduct a randomized controlled trial single-blind (examiner). The investigators included female patients diagnosed of fibromyalgia according to the American College of Rheumatology (ACR).

Thirty-four women with fibromyalgia are included and randomized into 2 groups: telerehabilitation program group based on aerobic exercise and control group. Exercise group receive 2 treatment sessions a week over 15 weeks.

All the variables are measured at the beginning of intervention and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed medically with Fibromyalgia
* Diagnosed according to the American College of Rheumatology criteria
* Age between 30 and 75 years old
* Telerehabilitation equipment including a laptop computer and access to internet

Exclusion Criteria:

* Any kind of contraindications for physical activity
* Other physical or psychological therapies in the last 3 months.
* Medication modifications in the last 3 months

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline
  The investigators measure the intensity of pain with a Visual Analogic Scale at baseline. The scale score ranges from 0 to 100 and higher scores indicate greater pain intensity.
Pain Intensity | Post-intervention, an average 15 weeks
  The investigators measure the intensity of pain with a Visual Analogic Scale (VAS) at the end of the intervention. The scale score ranges from 0 to 100 and higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Impact of fibromyalgia (Fibromyalgia Impact Questionnaire) | Baseline
  The investigators measure the impact of fibromyalgia with the Fibromyalgia Impact Questionnaire at baseline
Impact of fibromyalgia (Fibromyalgia Impact Questionnaire) | Post-intervention, an average 15 weeks
  The investigators measure the impact of fibromyalgia with the Fibromyalgia Impact Questionnaire at post-intervention
Mechanical pain sensitivity | Baseline
  The investigators measure mechanical pain sensitivity of the 18 points described initially by the American College of rheumatology with an algometer at baseline
Pressure Pain Threshold | Post-intervention, an average 15 weeks
  The investigators measure mechanical pain sensitivity of the 18 points described initially by the American College of rheumatology with an algometer at the end of treatment
Pain Catastrophizing | Baseline
  The investigators measure the pain catastrophizing with the Pain Catastrophizing Scale at baseline. Total values range from 0 to 52 points. Higher values indicate a higher level of pain catastrophizing.
Pain Catastrophizing | Post-intervention, an average 15 weeks
  The investigators measure the pain catastrophizing with the Pain Catastrophizing Scale at post-intervention. Total values range from 0 to 52 points. Higher values indicate a higher level of pain catastrophizing.
Psychological distress | Baseline
  The investigators measure psychological distress levels with the Hospital Anxiety and Depression Scale at baseline.The questionnaire consists of two subscales and each subscale has a total score of 21 points. Higher scores represent higher levels of anxiety.
Psychological distress | Post-intervention, an average 15 weeks
  The investigators measure psychological distress levels with the Hospital Anxiety and Depression Scale (HADS) at post-intervention. The questionnaire consists of two subscales and each subscale has a total score of 21 points. Higher scores represent higher levels of anxiety.
Upper limb function | Baseline
  The investigators measure upper limb functional capacity with the the Arm Curl Test at baseline. The number of repetitions that the participant can flex and re-extend the elbow holding a weight in 30 seconds is recorded.
Upper limb function | Post-intervention, an average 15 weeks
  The investigators measure upper limb functional capacity with the Arm Curl Test at post-intervention. The number of repetitions that the participant can flex and re-extend the elbow holding a weight in 30 seconds is recorded.
Lower limb function | Baseline
  The investigators measure lower limb functional capacity with the 6-Minute Walk Test at baseline. The distance (meters) that the patient can walk in 6 minutes is recorded.
Lower limb function | Post-intervention, an average 15 weeks
  The investigators measure lower limb functional capacity with the 6-Minute Walk Test at post-intervention. The distance (meters) that the patient can walk in 6 minutes is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Hernando, PT, Principal Investigator — University of Valladolid
Locations (1):
- Health Sciences Faculty, University of Valladolid, Soria, Spain

IPD SHARING:
Plan to Share IPD: No
The patient data were confidential and were assigned a number to each patient to maintain confidentiality